CLINICAL TRIAL: NCT00004354
Title: Study of Prevalence and Clinical Phenotype in Patients With Glucocorticoid-Remediable Aldosteronism
Status: Completed | Type: Observational
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Brigham and Women's Hospital (Other)
Other Study IDs: 199/11917; BWH-91328603
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-05

CONDITIONS: Hyperaldosteronism
Keywords: endocrine disorders; genetic diseases and dysmorphic syndromes; hyperaldosteronism; rare disease
MeSH Terms: conditions — Hyperaldosteronism; Endocrine System Diseases; Genetic Diseases, Inborn; Rare Diseases

SUMMARY:
OBJECTIVES: I. Determine the prevalence of glucocorticoid-remediable aldosteronism (GRA) in various hypertensive populations and screen at risk members of GRA pedigrees.

II. Investigate other factors regulating blood pressure in GRA (environmental, genetically determined factors).

III. Investigate renal and hormonal mechanisms regulating potassium homeostasis in GRA.

IV. Describe clinical phenotype of GRA patients. V. Prospectively screen GRA-affected patients with MRI angiography for intracranial aneurysm.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

Patients are screened for high blood pressure, suppressed plasma renin activity level, and low potassium levels. Urine is collected for a 24 hour period. Blood specimen is collected for molecular biologic evaluation for the presence of the chimeric gene diagnostic of GRA. Any history of cardiovascular events is recorded.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Diagnosed glucocorticoid-remediable aldosteronism (GRA) with hypertension Hypokalemia is variably seen Blood pressure variably elevated Elevated level of aldosterone Low level of plasma renin activity

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-06

CONTACTS AND LOCATIONS:
Overall Officials: Robert G. Dluhy, Study Chair — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States